CLINICAL TRIAL: NCT02392494
Title: A Single Rising Dose Study to Evaluate Safety, Pharmacokinetics and Pharmacodynamics of MK-1075 in HCV-Infected Patients
Brief Title: Evaluation of MK-1075 in Participants With Hepatitis C Virus (HCV) Infection (MK-1075-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1075-002; 2015-000127-93 (EudraCT Number); MK-1075-002 (Other: Merck Protocol Number)
Record Dates: First submitted 2015-03-16; First posted 2015-03-19 (Estimated); Results first posted 2018-12-31 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Intervention Model Description: In each panel (A, B, C, and D), participants will receive a single dose of MK-1075 (100, 200, 400, and 800 mg, respectively) in a fasted state. Safety and viral load (VL) data from the previous panel will be assessed before dosing the subsequent panel.
Oversight: Data Monitoring Committee: No

ARMS (4):
- MK-1075 100 mg (Panel A) (Experimental): HCV-infected participants receive a single 100 mg dose of MK-1075.
  Interventions: Drug: MK-1075
- MK-1075 200 mg (Panel B) (Experimental): HCV-infected participants receive a single 200 mg dose of MK-1075.
  Interventions: Drug: MK-1075
- MK-1075 400 mg (Panel C) (Experimental): HCV-infected participants receive a single 400 mg dose of MK-1075.
  Interventions: Drug: MK-1075
- MK-1075 800 mg (Panel D) (Experimental): HCV-infected participants receive a single 800 mg dose of MK-1075.
  Interventions: Drug: MK-1075

INTERVENTIONS:
Drug: MK-1075 — MK-1075 supplied as 10 mg or 100 mg tablets for oral administration.

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetics of MK-1075, and to determine the ability of MK-1075 to reduce HCV viral load, following administration of a single dose in HCV-infected participants.

DETAILED DESCRIPTION:
Per protocol, panels may be omitted if the objectives of the study are met in preceding panels.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of non-child bearing potential
* In good health other than HCV genotype (GT) 1 infection

Exclusion Criteria:

* Is mentally incapacitated or legally institutionalized
* Has a history of clinically significant and not stably controlled endocrine, gastrointestinal, cardiovascular, hematological, hepatic (excepting HCV infection), immunological, renal, respiratory, genitourinary or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Has a history of cancer
* Is positive for hepatitis B surface antigen (HBsAg) or human immunodeficiency virus (HIV)
* Has participated in another investigational trial within 4 weeks (or 5 half-lives) prior to Screening
* Consumes >2 alcoholic beverages a day or uses illegal drugs
* Has evidence or history of chronic hepatitis not caused by HCV including but not limited to non-HCV viral hepatitis, non-alcoholic steatohepatitis (NASH), drug-induced hepatitis, or autoimmune hepatitis
* Has clinical or laboratory evidence of advanced or decompensated liver disease, evidence of bridging fibrosis or higher grade fibrosis (Metavir score ≥3) from prior liver biopsy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2015-08-10 (Actual); Study Completion 2015-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Nine participants were enrolled and allocated to single doses of either 100, 200, or 400 mg of MK-1075. As per the protocol, planned Panel D (800 mg MK-1075) was not enrolled since the study objective was achieved in Panel C.
Groups:
- MK-1075 800 mg (Panel D): HCV-infected participants were to receive a single 800 mg dose of MK-1075. No participants were enrolled in this arm.
Period: Overall Study
Arm/Group | MK-1075 100 mg (Panel A) | MK-1075 200 mg (Panel B) | MK-1075 400 mg (Panel C) | MK-1075 800 mg (Panel D)
Started | 3 | 3 | 3 | 0
Completed | 3 | 3 | 3 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-1075 100 mg (Panel A) | MK-1075 200 mg (Panel B) | MK-1075 400 mg (Panel C) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (15.7) | 44.0 (8.0) | 49.7 (2.5) | 47.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 3
  Male | 1 | 3 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of the Sponsor's product, was also an AE. The percentage of participants that experienced an AE was reported for each treatment panel.
Time Frame: Up to Study Day 14
Population: All Participants as Treated (APaT): all participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-1075 100 mg (Panel A) | MK-1075 200 mg (Panel B) | MK-1075 400 mg (Panel C)
Number analyzed (Participants) | 3 | 3 | 3
Percentage of Participants | 66.7 | 66.7 | 33.3

2. Primary Outcome: Percentage of Participants Who Discontinued Study Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of the Sponsor's product, was also an AE. The percentage of participants that discontinued the study due to an AE was reported for each treatment panel.
Time Frame: Up to Study Day 14
Population: APaT: all participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-1075 100 mg (Panel A) | MK-1075 200 mg (Panel B) | MK-1075 400 mg (Panel C)
Number analyzed (Participants) | 3 | 3 | 3
Percentage of Participants | 0 | 0 | 0

3. Primary Outcome: Maximum HCV Viral Load (VL) Change From Baseline Over Time Following Single-Dose MK-1075
Description: For assessment of antiviral activity of MK-1075 at each study dose, baseline and post-dose HCV ribonucleic acid (RNA) (log10) were measured at pre-dose and 2, 4, 8, 12, 16, 24, 32, 48, 72, and 120 hours post-dose. For each participant, baseline measurement was defined as the measurement obtained pre-dose on the first day of dosing. The estimated change from baseline in HCV RNA VL (log10) was calculated for each participant by time point after each single dose, and the maximum change (reduction) in HCV RNA was determined and reported for each treatment arm using an Analysis of Variance (ANOVA) model.
Time Frame: Pre-dose (baseline), 2, 4, 8, 12, 16, 24, 32, 48, 72, and 120 hours post-dose
Population: Per Protocol (PP) Population: all participants who received at least 1 dose of study drug and who complied with the protocol
Measure: Mean (Standard Error); unit: log(IU/ml)
Arm/Group | MK-1075 100 mg (Panel A) | MK-1075 200 mg (Panel B) | MK-1075 400 mg (Panel C)
Number analyzed (Participants) | 3 | 3 | 3
log(IU/ml)
  Baseline HCV RNA | 5.72 (0.016) | 6.837 (0.145) | 6.31 (0.336)
  Maximum HCV RNA Change | 0.673 (0.078) | 1.15 (0.315) | 1.593 (0.134)

ADVERSE EVENTS:
Time Frame: Up to study day 14
Description: APaT: all participants who received at least 1 dose of study drug.
Arm/Group | MK-1075 100 mg (Panel A) | MK-1075 200 mg (Panel B) | MK-1075 400 mg (Panel C)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-1075 100 mg (Panel A) (N=3) | MK-1075 200 mg (Panel B) (N=3) | MK-1075 400 mg (Panel C) (N=3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.